CLINICAL TRIAL: NCT04552431
Title: Ciprofloxacin or Tamsulosin in Men With Chronic Prostatitis/Chronic Pelvic Pain Syndrome: a Randomized, Double-blind Trial
Brief Title: Chronic Prostatitis Collaborative Research Network Clinical Trial- Ciprofloxacin and Tamsulosin
Acronym: CPCRN RCT1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CPCRN RCT1; U01DK065209 (NIH)
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Prostatitis | interventions — Ciprofloxacin; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Men assigned to placebo
  Interventions: Drug: Tamsulosin Hydrochloride Placebo; Drug: Ciprofloxacin placebo
- Ciprofloxacin alone (Experimental): Men assigned to Ciprofloxacin alone
  Interventions: Drug: Ciprofloxacin; Drug: Tamsulosin Hydrochloride Placebo
- Tamsulosin alone (Experimental): Men assigned to Tamsulosin alone
  Interventions: Drug: Tamsulosin Hydrochloride; Drug: Ciprofloxacin placebo
- Combination of ciprofloxacin and tamsulosin (Experimental): Men assigned to a combination of ciprofloxacin and tamsulosin
  Interventions: Drug: Ciprofloxacin; Drug: Tamsulosin Hydrochloride

INTERVENTIONS:
Drug: Ciprofloxacin — Ciprofloxacin, 500 mg twice daily
  Other Names: CF
  Arms: Ciprofloxacin alone; Combination of ciprofloxacin and tamsulosin
Drug: Tamsulosin Hydrochloride — Tamsulosin Hydrochloride, 0.4 mg once daily
  Other Names: TH
  Arms: Combination of ciprofloxacin and tamsulosin; Tamsulosin alone
Drug: Tamsulosin Hydrochloride Placebo — Tamsulosin Hydrochloride Placebo (Placebo-TH) one tablet once daily
  Other Names: Placebo-TH
  Arms: Ciprofloxacin alone; Placebo
Drug: Ciprofloxacin placebo — Ciprofloxacin placebo (Placebo-CF) one tablet twice daily
  Other Names: Placebo-CF
  Arms: Placebo; Tamsulosin alone

SUMMARY:
Although the cause of chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) is unknown, physicians sometimes try to treat it with antibiotics or alpha-receptor blockers.

In this multicenter, double-blind factorial trial, 196 men with moderately severe CP/CPPS were randomly assigned to 6 weeks of treatment with ciprofloxacin, tamsulosin, both drugs, or placebo. Neither ciprofloxacin nor tamsulosin substantively reduced symptoms.

Ciprofloxacin and tamsulosin were not effective treatments for CP/CPPS. Patients had long-standing, refractory CP/CPPS and received trial treatments for only 6 weeks. Patients with new diagnoses who are given longer courses of the trial treatments might respond differently.

DETAILED DESCRIPTION:
Chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) is a common disorder and accounts for approximately 2 million visits to physicians annually in the United States. The substantial impact of CP/CPPS includes bothersome lower urinary tract symptoms, sexual dysfunction, reduced quality of life, and increased health care expenditures. The syndrome is diagnosed only on the basis of symptoms, principally pain or discomfort in the pelvic region. No objective measures can help define the disease. Although bacteria can infect the prostate, most men with prostatitis have a negative midstream urine culture, indicating that bacteria may not be the cause of their symptoms. Such men are classified as having National Institutes of Health (NIH) category III prostatitis, the most common of the clinically defined prostatitis syndromes. It is by no means clear that the disease is characterized by inflammation of the prostate or that the prostate is responsible for symptoms in a substantial proportion of patients. Because of this uncertainty, the term CP/CPPS is used. Chronic prostatitis/chronic pelvic pain syndrome is commonly seen by primary care practitioners, internists, and urologists. In the Olmsted County Study of Urinary Symptoms and Health Status Among Men, a population-based study in Olmstead County, Minnesota, the overall prevalence rate of a physician-assigned diagnosis of prostatitis was 9%. Population-based surveys of symptoms have estimated that the prevalence of the syndrome ranges from 9% to 12% among men. It is difficult to estimate the proportion of patients with symptoms lasting longer than 3 months whose disorder remains refractory to empirical therapy. These patients are commonly seen by urologists, but whether they represent a minor subpopulation of the overall symptomatic group or make up the majority of patients is unknown. The investigators chose to study these patients because they present with a troubling, long-standing problem and are usually treated with agents of unclear benefit. Even if a relatively large number of men whose symptoms last 3 months or more are cured by standard empirical therapy and the clinical scenario the investigators describe is uncommon, men with refractory symptoms still present a substantial problem to internists and urologists who have little information to guide therapy. Because the cause of CP/CPPS is unknown, affected men receive many empirical therapies. The 2 most common treatments prescribed by physicians are antimicrobial agents and alpha-adrenergic receptor antagonists, although there is little objective evidence to support their use. Quinolones, such as ciprofloxacin, are commonly used to treat CP/CPPS because of their excellent penetration into the prostate and broad spectrum of coverage for uropathogens and other organisms traditionally believed to be associated with the syndrome. Tamsulosin, an alpha-blocker, is an effective treatment for lower urinary tract symptoms in men with benign prostatic hyperplasia, and it has been hypothesized that tamsulosin may improve these symptoms in men with CP/CPPS. This randomized clinical trial was designed to evaluate whether ciprofloxacin or tamsulosin reduces symptoms of long-standing CP/CPPS of at least moderate severity, typical of the 488 men in our Chronic Prostatitis Cohort Study. The primary purpose of the trial was to test the most common prescription treatments given to men with CP/CPPS, who are commonly seen in our referral-based urologic practices.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of men with symptoms of discomfort or pain in the pelvic region for at least a 3-month period within the previous 6 months. Candidates must have at least a "moderate" overall score on the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI), defined as 15 or more points of a potential of 0 to 43 points.

Exclusion Criteria:

* Medical History and Comorbid Conditions: Prostate, bladder, or urethral cancer, seizure disorder. Concurrent history of Inflammatory bowel disease; active urethral stricture; neurologic disease or disorder affecting the bladder; liver disease; neurologic impairment or psychiatric disorder preventing understanding of consent and ability to comply with protocol. Diagnosed with or treated for symptomatic genital herpes in the prior 12 months.
* Urinary tract infection, with a urine culture value of greater than 100,000 colony forming units (CFU)/mL; clinical evidence of urethritis, including urethral discharge or positive culture, diagnostic of sexually transmitted diseases (including gonorrhea, chlamydia, mycoplasma or trichomonas, but not including HIV/AIDS); symptoms of acute or chronic epididymitis in the prior 3 months.
* Prior Treatment: Pelvic radiation, systemic chemotherapy; intravesical chemotherapy; intravesical Bacillus Calmette-Guerin (BCG), transurethral resection of the prostate (TURP), transurethral incision of the prostate (TUIP), transurethral Incision or Resection of the Bladder Neck (TUIBN), transurethral microwave therapy (TUMT), transurethral needle ablation (TUNA), balloon dilation of the prostate, open prostatectomy or any other prostate surgery or treatment such as cryotherapy or thermal therapy; prior treatment for orchialgia without pelvic symptoms; known allergy or sensitivity to ciprofloxacin hydrochloride, tamsulosin hydrochloride, or any of their known components. Prostate biopsy in the prior 3 months.
* Prior or Concurrent Medications: Concurrent use of Theophylline; on-going use of magnesium, aluminum, or calcium-containing antacids. Initiated or stopped finasteride or other androgen hormone inhibitors in the prior 6 months. Tamsulosin hydrochloride, doxazosin mesylate, terazosin HCl, or alpha-blockers; ciprofloxacin hydrochloride; antimicrobial agents (oral or parenteral); started, stopped, or changed dose level of any prostatitis-specific medications in the prior 4 weeks.
* Bioflavonoid agents; zinc or iron supplements; cimetidine in the prior 2 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 1997-09-30 (Actual); Primary Completion 2003-08-31 (Actual); Study Completion 2003-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the NIH-CPSI total score | Baseline and 6 weeks
  Change in the overall NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) total score (range of 0-43 points) from baseline to 6 weeks; a higher score indicates a worse outcome

SECONDARY OUTCOMES:
Change in the 7-point patient-reported global response assessment (GRA) | 6 weeks
  GRA assesses the change in overall symptoms from baseline to 6 weeks using a 7-point scale which ranges from:(0) markedly worse to (6) markedly improved.
Change in the physical summary scores on the Medical Outcomes Study 12-Item Short-Form Health Survey (MOS SF-12) | Baseline and 6 weeks
  Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP).
Change in the mental summary scores on the Medical Outcomes Study 12-Item Short-Form Health Survey (MOS SF-12) | Baseline and 6 weeks
  Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH).
Change in the pain scores of the NIH-CPSI | Baseline and 6 weeks
  Change in the pain scores of the NIH-CPSI (range of 0-21 points) from baseline to 6 weeks; a higher score indicates a worse outcome
Change in the voiding scores of the NIH-CPSI | Baseline and 6 weeks
  Change in the voiding scores of the NIH-CPSI (range of 0-10 points) from baseline to 6 weeks; a higher score indicates a worse outcome
Change in the quality of life scores of the NIH-CPSI | Baseline and 6 weeks
  Change in the quality of life scores of the NIH-CPSI (range of 0-12 points) from baseline to 6 weeks; a higher score indicates a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Landis, Principal Investigator — UNIVERSITY OF PENNSYLVANIA, PHILADELPHIA

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository: https://repository.niddk.nih.gov/home/
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- [Background] Propert KJ, Alexander RB, Nickel JC, Kusek JW, Litwin MS, Landis JR, Nyberg LM, Schaeffer AJ; Chronic Prostatitis Collaborative Research Network. Design of a multicenter randomized clinical trial for chronic prostatitis/chronic pelvic pain syndrome. Urology. 2002 Jun;59(6):870-6. doi: 10.1016/s0090-4295(02)01601-1. PMID 12031372